CLINICAL TRIAL: NCT00351806
Title: AISTCM-The Pathological Pattern Differentiation and Outcome Measurement of Acute Ischemic Stroke Treated With Traditional Chinese Medicine
Brief Title: AISTCM-Outcome Measurement of Acute Ischemic Stroke With Traditional Chinese Medicine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2004BA721A02
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Cerebral Infarction
Keywords: acute intracerebral infarction
MeSH Terms: conditions — Cerebral Infarction

ARMS (2):
- Chinese herbal medicine (Experimental)
  Interventions: Drug: Erigeron breviscapus injection; Drug: hua tuo zai zao wan (a herbal medicine pill); Drug: Compound stroke herbal medicine (8 herbal)
- placebo (Placebo Comparator)

INTERVENTIONS:
Drug: Erigeron breviscapus injection
  Arms: Chinese herbal medicine
Drug: hua tuo zai zao wan (a herbal medicine pill)
  Arms: Chinese herbal medicine
Drug: Compound stroke herbal medicine (8 herbal)
  Arms: Chinese herbal medicine

SUMMARY:
The purpose of this study is to determine whether Traditional Chinese Medicine (TCM) is able to improve the outcome of acute ischemic stroke and to observe its safety.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether Traditional Chinese Medicine (TCM) is able to improve the outcome of acute ischemic stroke and safety.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke diagnosis by CT/MRI scan
* Yin pattern of Traditional Chinese Medicine Theory
* 40-85 years old
* Total anterior circulation infarcts (TACI), partial anterior territory cerebral infarction (PACI), lacunar anterior circulation infarcts (LACI) type under Oxfordshire Community Stroke Project (OCSP) standard
* NIHSS >=4;
* Glasgow coma scale (GCS) >=7;
* Modified Rankin Scale less than 2 degrees before onset of this stroke
* Informed consent signed by patient or his/her family

Exclusion Criteria:

* Hemorrhagic stroke;
* Coma, GCS<=7;
* Cerebral hernia;
* Serious heart, liver, lung, kidney functional failure;
* Gastrointestinal (GI) bleeding;
* Thrombolysis drugs or surgery was administrated to the patient;
* Not cooperative with physician;
* Psychological disorder;
* Already taken part in other clinical drug trial within the past 3 months

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2005-07; Study Completion 2006-11

PRIMARY OUTCOMES:
death rate, Barthel Index

SECONDARY OUTCOMES:
Glasgow Outcome Scale (GOS)
Modified Rankin Scale (mRS)
National Institute of Health Stroke Scale (NIHSS)
Stroke Specific Quality of Life (SSQOL)
Scale of Traditional Chinese Medicine (SSTCM)

CONTACTS AND LOCATIONS:
Overall Officials: Longhui Yang, Chairmam, Study Chair — Branch of Science and Education
Locations (22):
- China (22):
  - Dongzhimen Hospital of Beijing University of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - Foshan Hospital of Traditional Chinese Medicine, Foshan, Guangdong
  - 2nd hospital of Zhongshan University, Guangzhou, Guangdong
  - Neurology Center, Guangdong Province Hospital of Tradtional Chinese Medicine, Guangzhou, Guangdong
  - Zhongshan Hospital of Traditional Chinese Medicine, Zhongshan, Guangdong
  - Ruikang Hospital of Traditional Chinese Medicine, Nanning, Guangxi
  - 1st Hospital of Guangxi college of Traditional Chinese Medicine, Nanning, Guangxi
  - The 1st Hospital of He'nan College of Traditional Chinese Medicine, Zhengzhou, Henan
  - The teahing hospital of Hubei College of Traditional Chinese Medicine, Wuhan, Hubei
  - Taizhou Hospital of Traditional Chinese Medicine, Taizhou, Jiangsu
  - Jinan Hospital of Traditional Chinese Medicine, Jinan, Shandong
  - Longhua Hospital of Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shanghai Hospital of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shuguang Hospital of Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Yueyang Hospital of Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - zhongshan hospital of Fudan Unversity, Shanghai, Shanghai Municipality
  - Huashan Hospital of Fudan Unveristy, Shanghai, Shanghai Municipality
  - The Hosptial of Shanxi College of Traditional Chinese Medicine, Xian Yang, Shanxi
  - The People's Hospital of Sichuan Province, Chengdu, Sichuan
  - Xinjiang Uygur Autonomous Region Hospital of Traditional Chinese Medicine, Ürümqi, Xinjiang
  - Zhejiang Province Hospital of Traditional Chinese Medicine, Hangzhou, Zhejiang
  - The 2nd Hospital of Wenzhou Medical College, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Huang Y, Guo JW; Project Group for Demonstration Study of Syndrome Differentiation Protocol and Effect Evaluation of Acute Ischemic Stroke. Outcome and safety assessment of an herbal medicine treatment protocol for yin pattern of acute ischemic stroke. Zhong Xi Yi Jie He Xue Bao. 2010 May;8(5):417-26. doi: 10.3736/jcim20100504. PMID 20456839